CLINICAL TRIAL: NCT03058432
Title: Concurrent Chemotherapy for Elderly Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-2016-HN03
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy; Chemoradiotherapy

STUDY DESIGN:
Intervention Model Description: Concurrent cisplatin based chemoradiotherapy versus radiotherapy alone

ARMS (2):
- Intensity-modulated Radiotherapy (Experimental): Radiotherapy alone was given.
  Interventions: Radiation: Radiotherapy alone
- Concurrent chemoradiotherapy (Active Comparator): Concurrent cisplatin-based radiotherapy was given.
  Interventions: Radiation: Concurrent chemoradiotherapy

INTERVENTIONS:
Radiation: Radiotherapy alone
  Arms: Intensity-modulated Radiotherapy
Radiation: Concurrent chemoradiotherapy
  Arms: Concurrent chemoradiotherapy

SUMMARY:
Concurrent Chemotherapy for Elderly Patients With Locoregionally Advanced Nasopharyngeal Carcinoma

DETAILED DESCRIPTION:
To evaluate concurrent chemotherapy for elderly patients with locoregionally advanced nasopharyngeal carcinoma treated by intensity-modulated radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated and histologically confirmed locoregionally advanced nasopharyngeal carcinoma

Exclusion Criteria:

* A history of another invasive cancer, prior RT to the head and neck area, prior cytotoxic chemotherapy or anti-EGFR therapy or the presence of any serious medical conditions,supposed to live less than 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
therapeutic success | From date of treatment until the date of completing treatment 1 month later
  A combined primary end point, named "therapeutic success"(TS), was used; it took into account activity, toxicity, and compliance.A TS was defined as a patient completing radiotherapy at the planned dose and schedule (no re-treatment delays beyond 2 weeks), and having an objective response (either complete or partial based on RECIST criteria) without (1) grade 3-4 nonhematological toxicity, (2) complications associated with hematologic toxicity such as febrile neutropenia, infection, bleeding, or transfusion, or (3) any toxicity leading to hospitalization or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaozhong Chen, Hangzhou, Zhejiang, China